CLINICAL TRIAL: NCT06316414
Title: Effects of Omalizumab on Food Allergy in Children With Severe Asthma: A Real Life Study
Brief Title: Omalizumab in Severe Asthmatics With Food Allergy
Acronym: OSAFA
Status: Completed | Type: Observational
Sponsor: Bambino Gesù Hospital and Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 1501/17
Record Dates: First submitted 2024-03-06; First posted 2024-03-18 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Food; Allergy, Anaphylactic Shock; Asthma in Children
MeSH Terms: conditions — Hypersensitivity; Anaphylaxis | interventions — Omalizumab

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes

GROUPS / COHORTS (1):
- Severe asthmatics with history of food anaphylaxis: Omalizumab will be administered i.m. with doses ranging from 150 mg every 28 days to 600 mg every 14 days, according to EMA dosing range table.
  Interventions: Biological: Omalizumab

INTERVENTIONS:
Biological: Omalizumab — Administration of Omalizumab at the doses indicated for asthma in the EMA information leaflet.

SUMMARY:
A prospective assessment of the impact of Omalizumab in terms of efficacy, safety, and quality of life (FA-QoL) in patients with moderate/severe asthma and history of anaphylaxis to peanut, tree nuts, fish, egg, milk, and/or wheat. Evaluation of the trend of total and specific IgE during Omalizumab treatment.

DETAILED DESCRIPTION:
Children (6-18 yrs) with severe asthma eligible for treatment with Omalizumab and reporting food anaphylaxis to be assessed for their concomitant food allergy.

At T0:

* oral food challenges (OFCs) to establish the threshold of reaction to the culprit food(s);
* number and severity of food-allergic reactions in the previous 12 months recorded
* Asthma Control Test
* Food Allergy-Quality of Life (FA-QoL) questionnaire
* total IgE
* specific IgE for the culprit foods

At T1 - four months after starting Omalizumab treatment:

* OFCs to the previously positive foods with evaluation of the threshold of reaction
* number and severity of food-allergic reactions in the previous 4 months recorded
* Asthma Control Test
* Food Allergy-Quality of Life (FA-QoL) questionnaire
* total IgE
* specific IgE for the culprit foods

At T2 - eight months after starting Omalizumab treatment:

* OFCs to the previously positive foods with evaluation of the threshold of reaction
* number and severity of food-allergic reactions in the previous 4 months recorded
* Asthma Control Test
* Food Allergy-Quality of Life (FA-QoL) questionnaire
* total IgE
* specific IgE for the culprit foods

At T1 - twelve months after starting Omalizumab treatment:

* OFCs to the previously positive foods with evaluation of the threshold of reaction
* number and severity of food-allergic reactions in the previous 4 months recorded
* Asthma Control Test
* Food Allergy-Quality of Life (FA-QoL) questionnaire
* total IgE
* specific IgE for the culprit foods

ELIGIBILITY:
Inclusion Criteria:

* Age 6 - 18 years
* Severe persistent allergic asthma according to the GINA guidelines
* Sensitized to a perennial aeroallergen, as witnessed by positive skin test and/or in vitro reactivity
* Symptoms inadequately controlled with inhaled corticosteroids + another medication, as witnessed by an ACT ≤ 19
* On treatment with high dose inhaled corticosteroids + another medication. Threshold dose for inhaled corticosteroids set at 400 mcg/day budesonide (or equivalent doses) for children < 12 years, at 800 mcg/day for older patients.
* Immediate food allergy with anaphylactic symptoms within 1hr. of ingestion of milk, egg, wheat, peanut, hazelnut, and/or codfish.
* Total IgE < 70 and >1,500 kU/L at baseline
* Sensitivity to food allergen documented by a positive skin prick test result and/or allergen-specific IgE level, with 0.35 kU/L as a lower limit of eligibility
* Positive OFC within the past 12 months, with minimal or no reactions to the placebo challenge.
* Trained on the proper use of epinephrine
* In case of female subjects of child-bearing potential, negative human chorionic gonadotropin blood sample for pregnancy testing
* No known contraindications to oral immunotherapy with food protein or Omalizumab
* Parent/legal guardian written informed consent

Exclusion Criteria:

* Total IgE at screening > 70 or ≤ 2,500 kUI/L
* allergy to food(s) not investigated in this study
* Immune deficiency
* Previous reaction to Omalizumab
* Previous organ transplantation
* Use of monoclonal antibodies in the previous 6 months
* Subjects with gastrointestinal or gastroesophageal disease, chronic infections, scleroderma, hepatic and gallbladder disease, chronic non-allergic pulmonary disease.
* Subjects who have received an experimental drug in the last 30 days prior to admission into this study or who plan to use an experimental drug during the study
* Pregnant or breast-feeding females.
* Subjects with food protein induced enterocolitis syndrome (FPIES)
* Subjects is on a build-up phase of standard subcutaneous immunotherapy for inhalant allergens (may be enrolled on maintenance dose)
* Inability to discontinue antihistamines for 5 half-lives prior to routine study tests (OFC)
* Subjects with weight-IgE combination yielding a dose requirement greater than 600 mg according to the EMA schedule for Omalizumab
* Systemic steroids oral, IM, or IV for indications other than asthma for more than 3 weeks in the past 6 months.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: * Children with severe asthma eligible for treatment with Omalizumab consecutively enrolled at the Bambino Gesu Pediatrica Hospital IRCCS in Rome
  * ACT < 20
  * Food allergy as described
  * History of food-induced anaphylaxis
  * positive OFCs with milk, baked milk, egg, baked egg, wheat, peanut, hazelnut, codfish.
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Milligram tolerated food allergen (gms) of raw and baked milk, raw and baked egg, hazelnut, peanut, wheat, and/or fish at T1. | Four months (T1)
  Threshold of reactivity assessed as No Observed Adverse Events Level (NOAEL) to each of the analysed food

SECONDARY OUTCOMES:
Proportion of negative OFCs at T1 | Four months (T1)
  Percentage of OFC tolerated until the last dose of food.
NOAEL for raw and baked milk, raw and baked egg, hazelnut, peanut, wheat, and/or fish at T2. | Eight months (T2)
  Change in the NOAEL at the third OFC to the foods who did not pass the OFC at T1
NOAEL for raw and baked milk, raw and baked egg, hazelnut, peanut, wheat, and/or fish at T3. | Twelve months (T3)
  Change in the NOAEL at the fourth OFC to the foods who did not pass the OFC at T2
Change in number of anaphylactic events | Twelve months (T3)
  Number of episodes of anaphylaxis in the 6 - 12 months preceding T0 compared with those 6 - 12 months after the first dose of Omalizumab
Rate of severity of anaphylactic events | Twelve months (T3)
  Severity of episodes of anaphylaxis in the 6 - 12 months preceding T0 compared with those 6 - 12 months after the first dose of Omalizumab; PRACTALL score: 1 - mild, 2 - moderate, 3 - severe.
Asthma Control Test (ACT) | Twelve months (T3)
  Change from baseline in ACT score: 5 worse, 25 better outcome
Quality of Life score | Four (T1), eight (T2), twelve (T3) months
  Change from baseline in age-appropriate FA-QoL score: 0, better; 84, worse outcome
Total IgE | Four (T1), eight (T2), twelve (T3) months
  Change from baseline in total IgE
Specific IgE for milk, egg, hazelnut, peanut, wheat, and/or fish | Four (T1), eight (T2), twelve (T3) months
  Change from baseline in sIgE;

CONTACTS AND LOCATIONS:
Locations (1):
- Pediatric Hospital Bambino Gesù IRCCS - Allergy Dpt, Roma, Italy

IPD SHARING:
Plan to Share IPD: Yes
Anonymized Individual Participating Data will be made available to researchers upon reasonable request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data requests can be submitted starting 9 months after article publication and the data will be made accessible for up to 24 months. Extensions will be considered on a case-by-case basis.
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information or to submit a request, please contact alexfioc@gmail.com

REFERENCES:
- [Background] Fiocchi A, Artesani MC, Riccardi C, Mennini M, Pecora V, Fierro V, Calandrelli V, Dahdah L, Valluzzi RL. Impact of Omalizumab on Food Allergy in Patients Treated for Asthma: A Real-Life Study. J Allergy Clin Immunol Pract. 2019 Jul-Aug;7(6):1901-1909.e5. doi: 10.1016/j.jaip.2019.01.023. Epub 2019 Feb 20. PMID 30797778
- [Derived] Arasi S, Bitetti C, Lo Scalzo L, Spagnoli A, Fabrizi E, Fiocchi A, Cafarotti A. Omalizumab Dose-Related Efficacy in a Cohort of Children With Severe Food Allergy: OSAFA Observational Study. Allergy. 2026 Jan 19. doi: 10.1111/all.70228. Online ahead of print. PMID 41555682
- [Derived] Arasi S, Cafarotti A, Galletta F, Panetta V, Riccardi C, Calandrelli V, Fierro V, Dahdah L, Artesani MC, Valluzzi RL, Pecora V, Tallarico V, Dinardo G, Lo Scalzo L, Fiocchi A. Omalizumab reduces anaphylactic reactions and allows food introduction in food-allergic in children with severe asthma: An observational study. Allergy. 2025 Apr;80(4):1074-1085. doi: 10.1111/all.16314. Epub 2024 Sep 16. PMID 39282750